CLINICAL TRIAL: NCT03281590
Title: Stroke and Cerebrovascular Diseases Registry
Status: Completed | Type: Observational
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Other Study IDs: 17-281
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2021-10

CONDITIONS: Stroke; Acute Stroke; Acute Brain Injury; Ischemic Stroke; Hemorrhagic Stroke; Transient Ischemic Attack; Subarachnoid Hemorrhage; Cerebral Ischemia; Cerebral Infarction; Cerebral Stroke; Venous Sinus Thrombosis, Cranial
Keywords: identification; diagnosis; management; investigation; prevalence; incidence; quality of care; hospitalization; morbidity; disability
MeSH Terms: conditions — Stroke; Brain Injuries; Ischemic Stroke; Hemorrhagic Stroke; Ischemic Attack, Transient; Subarachnoid Hemorrhage; Brain Ischemia; Cerebral Infarction; Sinus Thrombosis, Intracranial; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with stroke: Patients with the Acute Brain injury, Transient Ischemic Attack, Acute and Chronic Ischemic and Hemorrhagic Stroke, Subarachnoid hemorrhage, and cerebral venous thrombosis from pre-hospitalization, hospitalization (in-patient) and post hospitalization (clinic) data
- Patients without stroke: Control subject who have the risk factors but never had stroke.

SUMMARY:
This is a single institutional registry database for the patients with stroke and cerebrovascular diseases. Stroke is the fifth leading cause of death in the United States. Despite extensive research, most of the patients die or suffer from varying degree of post-stroke disabilities due to neurologic deficits. This registry aims to understand the disease and examine the disease dynamics in the local community.

DETAILED DESCRIPTION:
Stroke is the fifth cause of all-cause mortality in US http://www.cdc.gov/stroke/facts.htm Early identification and treatment not only prevent mortality but also morbidity. Recent advancement in the imaging and diagnostic technique and novel therapeutic modalities has dramatically helped to downgrade stroke from the list of top mortality index in the last 3 years. However, studies determining factors which help predict stroke outcome are still underway and much work needs to be done in this direction. Many factors currently are used to predict stroke outcome with varying results, for e.g. NIHSS is a good predictor of stroke outcome at 3 months; however, the investigators need better predictors, outcome scales or outcome measures which are easy, reliable and has better specificity and sensitivity.

Acute Brain injury, Transient Ischemic Attack is a special category of a neurological condition wherein there is an impending devastating outcome if workup is not completed in a timely fashion. There is an urgent need to do investigations with high-risk patients to prevent stroke and further mortality and morbidity. The abcd2 score can help us to risk stratify the TIA and to predict the chances of stroke in this specific cohort. However, investigators need better identifiers than already present, to improve the patient changes in secondary prophylaxis of stroke prevention http://www.stroke.org/sites/default/files/resources/tia-abcd2-tool.pdf?docID

There is also some correlation of clinical and biochemical predictors in subarachnoid, cerebral venous thrombosis including Hunt and Hess, SAH score, WFNS-SAH grading among others with variable predictive quality. (Rosen et al; Neurocritical Care; April 2005, Volume 2, Issue 2, pp 110-118: Subarachnoid hemorrhage grading scales).

ELIGIBILITY:
Inclusion Criteria:

1. All patients with a diagnosis of Acute Brain injury, Transient Ischemic Attack, Acute and Chronic Ischemic and Hemorrhagic Stroke, Subarachnoid hemorrhage, and cerebral venous thrombosis seen in UNMH.
2. Age >1 years of age.

Exclusion Criteria:

1. Patients who don't have the diagnosis of Acute Brain injury, Transient Ischemic Attack, Acute and Chronic Ischemic and Hemorrhagic Stroke, Subarachnoid hemorrhage, and cerebral venous thrombosis.
2. Patients who have Epidural Hematoma, Subdural hematoma.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a final/discharge diagnosis of stroke or transient ischemic attack can be included into the Stroke Registry. This includes cases with a principal/primary or secondary diagnosis of:
  * Cerebral Infarction
  * Intracerebral Hemorrhage (non-traumatic)
  * Ischemic Stroke
  * Subarachnoid Hemorrhage (non-traumatic)
  * Transient Ischemic Attack (TIA)
  * Acute Brain Injury
  * Cerebral Venous Sinus Thrombosis
  The investigators will use the available EMR and databases to search for these patients using relevant ICD-9/10 codes.
Sampling Method: Non-Probability Sample
Enrollment: 4594 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Improvement or worsening in stroke signs/symptoms. | 1 year
  Prospective and retrospective analysis of patients with the acute brain injury, transient ischemic attack, acute and chronic ischemic and hemorrhagic stroke, subarachnoid hemorrhage, and cerebral venous thrombosis from pre-hospitalization, hospitalization (in-patient) and post hospitalization (clinic) data to determine factors which can predict stroke outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Torbey, MD, MPH, Study Chair — University of New Mexico; Atif Zafar, MD, Principal Investigator — University of New Mexico; Asad Ikram, MD, Study Director — University of New Mexico; Mudassir Farooqui, MD, MPH, Study Director — University of New Mexico
Locations (1):
- Department of Neurology, University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No